CLINICAL TRIAL: NCT06891326
Title: Efficacy and Safety of Transcranial Alternating Current Stimulation for Depression: a Multicenter Randomized Controlled Trial Study
Brief Title: Efficacy and Safety of tACS for Depression: a Multicenter RCT Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai Mental Health Center (Other); Shandong Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20240913
Record Dates: First submitted 2024-09-29; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-09

CONDITIONS: Depression Disorders
Keywords: tACS; depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Sham Comparator)
  Interventions: Device: sham transcranial Alternating Current Stimulation
- Treatment group (Active Comparator)
  Interventions: Device: active tACS

INTERVENTIONS:
Device: sham transcranial Alternating Current Stimulation — we use fade-in, short-stimulation, fade-out (FSF) stimulation pattern, with 60s-long fade-in/out periods, 2.0mA peak current at the beginning and the end of stimulation session
  Arms: Control group
Device: active tACS — The active tACS protocol lasted for 40 min of continuous sine-wave stimulation with the frequency of 10Hz and an amplitude ranging from 1.5mA to 2.0mA, adjusted according to the tolerability among individuals.
  Arms: Treatment group

SUMMARY:
Transcranial alternating current stimulation (tACS) is a promising non-invasive technique for major depression, because of its advantage of lower risks and expenses compared to other therapies such as deep brain stimulation, electroconvulsive therapy, and repetitive transcranial magnetic stimulation. Randomized controlled trials (RCTs) of depression treated by tACS have been conducted but provided limited and incongruous results. We designed a multi-center RCT to evaluate the efficacy and safety of tACS for depression.

Eligible participants will be patients diagnosed with depression (HDRS-17≥8), aged 18 to 65, and without other conditions that could interfere with the study. A total of 72 participants will be recruited from 4 clinic centers. Participants will be randomized 1:1 to active tACS or sham stimulation group. The study staff and the participants are blinded to the randomization results. Stimulating electrodes will be placed on the scalp corresponding to bilateral dorsolateral prefrontal cortex (DLPFC) using frequency of 10Hz and amplitude of 1.5 to 2.0 mA. The intervention will last for 4 weeks, containing 20 40-minute sessions in total. Another 4-week observation will be followed by the end of the intervention. Participants will receive assessments at baseline, 2 weeks, 4 weeks, 6 weeks, and 8 weeks after the study begins. Psychological scales are used for the evaluation of their mental and quality of life. Besides, electroencephalogram (EEG) recording and magnetic resonance imaging (MRI) scans will also be performed to quantitatively measure the neural activities as well as the functional connectivity changes within the depression-related circuits.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of depressive disorder;
2. Age ranges between 18 and 65 years;
3. HDRS-17 score equals to or above 8;
4. No medical history/Under stable antidepressant treatment in one month;

Exclusion Criteria:

1. Combination of other psychotic disorders and neurological diseases;
2. History of invasive brain surgeries;
3. Non-invasive neurostimulation treatments within 3 months;
4. Physical condition that may endanger patients' safety during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-09-08 (Estimated); Study Completion 2026-10-08 (Estimated)

PRIMARY OUTCOMES:
Clinical remission | 4 weeks after the intervention
  The primary endpoint is defined as the decreased scores of Hamilton Depression Scale-17 (HDRS-17) at the 4-week follow-up compared to baseline scores. HDRS ranges from 0 to 68, with higher scores indicating more severe depression symptoms. The two-sample t-test is used to test the difference in score changes between the treatment group and control group at the 4-week follow-up visit point.

SECONDARY OUTCOMES:
Adverse events | 8 weeks, when the study is completed
  The adverse events will be reported by physicians at the 8-week follow-up visit, which items include the number of the events, the severe levels of each event, and its duration time.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Ruijin Hospital affiliated to Shanghai JiaoTong University School of Medicine, Shanghai
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR